CLINICAL TRIAL: NCT06952023
Title: Pulsed Field-Based Bi-atrial Maze-like Catheter Ablation Versus Pulmonary Vein Isolation in Persistent Atrial Fibrillation: A Multi-center Randomized Controlled Trial
Brief Title: PFA-based Bi-atrial Maze-like Catheter Ablation for PeAF
Acronym: PEACE-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: maze001
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Desmoglein 1

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PF-based modified Maze ablation (Experimental): patients will receive PF energy based PVI, BOX ablation, LA anterior wall linear ablation from the right superior pulmonary vein to the mitral annulus (under sinus rhythm), MI ablation, linear ablation of the RA posterior wall (up to the superior vena cava and down towards the inferior vena cava according to the potential), and CTI ablation.
  Interventions: Procedure: Modified Maze ablation with PFA
- RF-based PVI only (Active Comparator): PVI only with PF energy
  Interventions: Procedure: PVI only with PFA

INTERVENTIONS:
Procedure: Modified Maze ablation with PFA — Modified Maze ablation with PFA
  Arms: PF-based modified Maze ablation
Procedure: PVI only with PFA — PVI only with PFA
  Arms: RF-based PVI only

SUMMARY:
In radiofrequency (RF) ablation of persistent atrial fibrillation (PeAF), the additional linear ablation beyond pulmonary vein isolation (PVI) does not yield an reduce atrial arrhythmias recurrences.The goal of this clinical trial is to evaluate the efficiency of pulsed filed (PF) energy-based bi-atrial modified Maze ablation vs PF energy-based PVI of PeAF.

The main questions it aims to answer are:

Does PF energy effectively perform linear ablation in the left atrium? Does PFA-based bi-atrial modified Maze ablation significantly improve the success rate of PeAF ablation compared with PFA-based PVI?

Patients with PeAF who meet the criteria and undergo catheter ablation will be randomly assigned to the study group (PF-based bi-atrial modified Maze ablation group) and control group (PF-based PVI only) in a 1:1 ratio. All patients will received a 7-d Holter at 3-,6-,9-,12-month after the ablation. The primary endpoint is the freedom from documented atrial arrhythmia (AF/AFL/AT lasting for over 30 seconds) recurrence monitored by ECG, 7-day ambulatory ECG, or equivalent cardiac monitoring from 4th to 12th month after the procedure without taking I/III AADs.

DETAILED DESCRIPTION:
Patients with PeAF who meet the criteria and undergo catheter ablation will be randomly assigned to the study group (PF-based bi-atrial modified Maze ablation group) and control group (PF-based PVI only) in a 1:1 ratio. In the study group, patients will receive PF energy based PVI, BOX ablation, LA anterior wall linear ablation from the right superior pulmonary vein to the mitral annulus (under sinus rhythm), MI ablation, linear ablation of the RA posterior wall (up to the superior vena cava and down towards the inferior vena cava according to the potential), and CTI ablation. The patients in the control group will received PVI only with PF energy. If the patients do not restore to sinus rhythm, they will receive electrical cardioversion.

All patients received guideline-directed standardized drug therapy, including anti-arrhythmic medications, postoperatively. Discontinuation of all anti-arrhythmic drugs after the blanking period. All patients will received a 7-d Holter at 3-,6-,9-,12-month after the ablation. The primary endpoint is the freedom from documented atrial arrhythmia (AF/AFL/AT lasting for over 30 seconds) recurrence monitored by ECG, 7-day ambulatory ECG, or equivalent cardiac monitoring from 4th to 12th month after the procedure without taking I/III AADs.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with symptomatic PeAF at 18-75 years old who are eligible for the PFA procedure, and have any the following documentation, within 180 days of randomization of either: i. A 24-hour continuous ECG recording (from any regulatory cleared rhythm monitoring device) confirming continuous AF, OR ii. Two ECGs (from any regulatory cleared rhythm monitoring device) showing continuous AF taken at least 7 days，OR iii. physician note of persistent continuous AF for > 7 days
* The duration of AF lasting ≥ 1 year

Exclusion Criteria:

* PaAF or PeAF with duration < 1 year
* has received catheter ablation procedure for AF or atrial septal defect repair before enrollment
* left atrial diameter ≥55 mm or thrombosis in the left atrium
* eGFR<30mL/min/1.73m2
* a history of cerebrovascular disease within the last three months (including stroke and transient ischemic attack)
* acute or severe systemic infection
* refused to participate in this trial; or those who have participated in other clinical drug trials within 3 months prior to enrollment
* congenital heart disease, thyroid dysfunction, severe hepatic insufficiency (Child-Pugh classification B-C), severe coagulation dysfunction (international normalized ratio > 1.5 or partial activated prothrombin time prolonged by ≥ 10 seconds, or plasma prothrombin time prolonged by ≥ 3 seconds, or fibrinogen ≤ 1.5 g/L), or active bleeding
* pregnant women, breastfeeding women or women who plan to become pregnant during the study period, those who have a positive pregnancy test result during the screening period
* life expectancy < 12 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial tachycardia during blanking period to Month 12 | during blanking period to Month 12
  freedom of occurrence ≥ 30 sec of Atrial Fibrillation (AF), Atrial Flutter (AFL), atrial Tachycardia (AT); or any electrical cardioversion or re-ablation for AF, AFL, or AT; or any Class I or III AAD use

SECONDARY OUTCOMES:
Acute Success - Isolation rate of attempted pulmonary veins and left atrial linear ablation | intraprocedure
  Isolation rate of attempted pulmonary veins and left atrial linear ablation
device or procedure-related Composite Adverse Events | day 0 to 12 months
  device or procedure-related Composite Adverse Events including Heart block, Myocardial infarction, Peripheral or organ thromboembolism, Stroke/ Cerebrovascular accident/Transient ischemic attack (TIA),Unresolved phrenic nerve palsy / paresis,Vascular access complications
procedure time | intraprocedure
  procedure time

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Jiangsu Provincial Hospital, Nanjing, Jiangsu
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The Affiliated Hospital Of Medical School Of Ningbo University, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sun Y, Dai S, Xiao X, Wang Z, Yu X, Ma C, Zhang R, Gao L, Xia Y, Yin X. Tailored bi-atrial linear ablation guided by electrophysiological mapping for persistent atrial fibrillation. BMC Cardiovasc Disord. 2024 Nov 20;24(1):658. doi: 10.1186/s12872-024-04332-w. PMID 39567904